CLINICAL TRIAL: NCT04374682
Title: Effectiveness of a Home Based Exercise Program on Temporomandibular Dysfunction Syndrome: A Pilot Study in a Tertiary Care Hospital.
Brief Title: Effectiveness of a Home Based Exercise Program on Temporomandibular Dysfunction Syndrome
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, safaa Mahran, Associate Proffesor, Assiut University
Other Study IDs: 17300389
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Temporomandibular Disorder
Keywords: Temporomandibular dysfunction; Exercise; treatment; pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: exercises — stretching exercises - physiotherapy modalities - self care instructions

SUMMARY:
patients with chronic refractory temporomandibular dysfunction were prescribed home exercise and were followed for 6 months. Pain , mouth opening and Fonseca's were done at day 1 and after 6 months of the study.

DETAILED DESCRIPTION:
Each patient was seen by the rheumatologist who did the following; Full history taking including special habits like chewing gums or biting nails, Pain level measured by visual analogue scale 100 (both at rest and during temporomandibular joint movement) Clinical Examination of the temporomandibular joint including localized tenderness and amount of mouth opening After that the patients were prescribed the rehabilitation program in the form of heat modalities and Transcutaneous electric nerve stimulation on the on the temporomandibular joint, given an individual demonstration of the home based exercises and were given a reminding handout.

The rehabilitation program consisted of the following exercises: lateral deviation, protrusion/retraction and mandibular opening.

Isometric cervical muscle strengthening exercises were also prescribed for the patients.

Assessment of the severity of temporomandibular joint affection using the Fonseca's questionnaire were done twice; the first at the entry point to the study and once again after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering painful temporomandibular joint

Exclusion Criteria:

* Patients with history of face trauma
* Patients with surgery at the temporomandibular joint
* Dental procedure in the last 6 months period
* Patients with rheumatic diseases

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with chronic Temporomandibular pain refractory to medical treatment
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale for pain during rest and on moving the jaw | 6 months
  visual analogue scale 0-100 with higher score indicating more pain.
mouth opening | 6 months
  Distance between the edges of central incisors was measured. Measures are compared pre and post exercises.
Fonseca's scale. | 6 months
  It is composed of 10 questions, which include checking for the presence of pain in temporomandibular joint, head, back, and while chewing, parafunctional habits, movement limitations, joint clicking, perception of malocclusion, and sensation of emotional stress. The volunteers were informed that the 10 questions should be answered with "yes", "no" and "sometimes" and that only one answer should be marked for each question. Scoring ranges between 0-50 with higher score indicating worse results.

CONTACTS AND LOCATIONS:
Overall Officials: Safaa A Mahran, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
studying the effectiveness of stretching exercises on chronic temporomandibular dysfunction syndrome refractory to medical treatment

REFERENCES:
- [Background] Eweka OM, Ogundana OM, Agbelusi GA. TEMPOROMANDIBULAR PAIN DYSFUNCTION SYNDROME IN PATIENTS ATTENDING LAGOS UNIVERSITY TEACHING HOSPITAL, LAGOS, NIGERIA. J West Afr Coll Surg. 2016 Jan-Mar;6(1):70-87. PMID 28344938
- [Background] Kato MT, Kogawa EM, Santos CN, Conti PC. TENS and low-level laser therapy in the management of temporomandibular disorders. J Appl Oral Sci. 2006 Apr;14(2):130-5. doi: 10.1590/s1678-77572006000200012. PMID 19089044
- [Background] Cascos-Romero J, Vazquez-Delgado E, Vazquez-Rodriguez E, Gay-Escoda C. The use of tricyclic antidepressants in the treatment of temporomandibular joint disorders: systematic review of the literature of the last 20 years. Med Oral Patol Oral Cir Bucal. 2009 Jan 1;14(1):E3-7. PMID 19114953
- [Background] Carvalho CM, de Lacerda JA, dos Santos Neto FP, Cangussu MC, Marques AM, Pinheiro AL. Wavelength effect in temporomandibular joint pain: a clinical experience. Lasers Med Sci. 2010 Mar;25(2):229-32. doi: 10.1007/s10103-009-0695-y. Epub 2009 Jun 30. PMID 19565312